CLINICAL TRIAL: NCT02750592
Title: An Open-label, Phase III, Study of Subcutaneous Secukinumab to Assess Efficacy, Safety and Tolerability at up to 52 Weeks in Japanese Patients With Active Ankylosing Spondylitis
Brief Title: Study of Efficacy and Safety of Secukinumab in Japanese Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457H1301
Record Dates: First submitted 2016-04-04; First posted 2016-04-25 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; secukinumab; AIN457H; SpondyloArthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — secukinumab; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- secukinumab 150mg (Experimental): A screening (SCR) epoch running 4-10 weeks before baseline (BSL) was used to assess eligibility followed by 52 weeks of treatment. The treatment periods consist of Treatment period 1 (BSL to Week 24) and Treatment period 2 (Week 24 to Week 52). After Week 52 follows a post-treatment follow-up until Week 60. A follow-up visit was done at 12 weeks after last study treatment administration for all patients, regardless of whether they completed the entire study as planned (Week 60) or discontinue prematurely.
  Interventions: Drug: Secukinumab 150 mg provided in 1.0 mL pre-filled syringes (PFSs) for sc injection.

INTERVENTIONS:
Drug: Secukinumab 150 mg provided in 1.0 mL pre-filled syringes (PFSs) for sc injection. — Baseline, 1, 2, 3, 4 week. After 4 week, administered every 4 weeks.

SUMMARY:
The purpose of this study was to assess the clinical efficacy, safety and tolerability of secukinumab subcutaneous injections up to 52 weeks in Japanese patients with active AS despite current or previous non-steroidal anti-inflammatory drugs (NSAIDs) and/or anti-tumor necrosis factor (TNF) α therapy. Efficacy and safety data were used to support the registration of secukinumab in Japan for the treatment of active AS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe AS with prior documented radiologic evidence (x-ray or radiologist's report) fulfilling the Modified New York criteria for AS with active AS assessed by BASDAI ≥ 4 (0-10) and spinal pain as measured by VAS≥ 4 cm (BASDAI question #2) at Baseline
* Patients should have been on NSAIDs at the highest recommended dose for at least 3 months prior to baseline with an inadequate response or failure to respond, or less than 3 months if therapy had to be withdrawn due to intolerance, toxicity or contraindications
* Patients who have been on a TNFα inhibitor (not more than one) must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months prior to baseline or have been intolerant to at least one administration of an anti-TNFα agent

Exclusion Criteria:

* Patients with total ankylosis of the spine
* Patients previously treated with any biological immunomodulating agents except for those targeting TNFα
* Active ongoing inflammatory diseases other than AS that might confound the evaluation of the benefit of secukinumab therapy, including inflammatory bowel disease or uveitis
* Known infection with HIV, hepatitis B or hepatitis C at screening or baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 patients were screened, and 30 patients (81.1%) completed the screening phase and entered Treatment Period
Pre-assignment Details: Seven patients were screening failures
Groups:
- Secukinumab 150mg: A screening (SCR) epoch ran 4-10 weeks before baseline (BSL) and was used to assess eligibility followed by 52 weeks of treatment. The treatment periods consisted of Treatment period 1 (BSL to Week 24) and Treatment period 2 (Week 24 to Week 52). After Week 52 there was a post-treatment follow-up until Week 60. A follow-up visit was done at 12 weeks after last study treatment administration for all patients, regardless of whether they completed the entire study as planned (Week 60) or discontinued prematurely.
Period: Overall Study
Arm/Group | Secukinumab 150mg
Started | 30
Completed | 25
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: The safety set included all patients who took at least one dose of study treatment during the treatment periods.
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.25)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 27
  >=65years | 3
  >=75 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 30
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of SpondyloArthritis International Society 20 Response (ASAS20)
Description: This table is ASAS20 response using non-responder imputation for FAS
  It assesses the efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline in Japanese patients with active AS based on the proportion of patients achieving an ASAS (Assessment of SpondyloArthritis International Society criteria) 20 response.
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of ≥ 20% and ≥ 1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥ 20% and ≥ 1 unit on a scale of 10 in the remaining domain
Time Frame: week 16
Population: Full analysis set (FAS): The FAS comprised of all patients who entered into the treatment periods.
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 21

2. Secondary Outcome: ASAS 40 Response Rate With Non-responder Imputation (NRI)
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the proportion of patients achieving an ASAS 40 response
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain
Time Frame: Week 16
Population: FAS
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 14

3. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity (BASDAI) 50 Response Rate
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the proportion of patients achieving Bath Ankylosing Spondylitis Disease Activity (BASDAI) 50 response
  The BASDAI 50 is defined as an improvement of at least 50% in the BASDAI compared to baseline
Time Frame: Week 16
Population: FAS
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 11

4. Secondary Outcome: Change in High Sensitivity C-Reactive Protein (hsCRP)
Description: hsCRP (mg/L) change from baseline using observed data with log e transformation
  The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the change from baseline of high sensitivity C-Reactive Protein (hsCRP)
  hsCRP is measured as a marker of inflammation from blood samples during the study
Time Frame: baseline, Week 16
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
mg/L | 0.247 [0.125 to 0.487]

5. Secondary Outcome: Number of Participants With ASAS 5/6 Response Criteria
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the proportion of patients meeting the ASAS 5/6 response criteria
  The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains
Time Frame: Week 16
Population: FAS
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 14

6. Secondary Outcome: Mean Change From Baseline in BASDAI From Baseline
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the change from baseline in total BASDAI
  The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS
  Each question (question 1 to 6) is scored from 0 to 10 (0 being no problem and 10 being the worst problem). To give each symptom equal weighting, the mean (average) of the two scores relating to morning stiffness (questions 5 and 6) is taken. The mean of questions 5 and 6 is added to the scores from questions 1-4. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score.
Time Frame: Baseline, week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
scores on a scale | -3.088 (2.0697)

7. Secondary Outcome: Change From Baseline in Short Form Health Survey Physical Component Summary (SF-36 PCS) Score
Description: SF-36 PCS, mean change from baseline:
  The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the change from baseline in Short Form Health Survey Physical Component Summary (SF-36 PCS)
  The SF-36 is an instrument to measure health-related quality of life among healthy patients and patients with acute and chronic conditions
  Score range is from 0 (no problems) to 100 (unable to perform the activity)
  SF-36 is a 36 item questionnaire which measures Quality of Life across eight domains, which are both physically and emotionally based. Two overall summary scores, the Physical Component Summary (PCS) and Mental Component Summary (MCS) can be computed. In this study, SF-36 PCS is used to assess improvement from baseline. There is no total overall score; scoring is computed for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score.
Time Frame: Baseline, week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
scores on a scale | 6.306 (8.0724)

8. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL)
  The ASQoL is a self-administered questionnaire designed to assess health-related quality of life in adult patients with Ankylosing Spondylitis. The ASQoL contains 18 items with a dichotomous yes/no response option. A single point is assigned for each "yes" response and no points for each "no" response resulting in overall scores that range from 0 (least severity) to 18 (highest severity)
Time Frame: Baseline, week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
scores on a scale | -3.40 (4.00)

9. Secondary Outcome: Proportion of Participants Achieving ASAS Partial Remission
Description: The efficacy of secukinumab 150 mg s.c. at Week 16 relative to baseline based on the proportion of patients achieving an ASAS partial remission
  The ASAS partial remission criteria are defined as a value not above 2 units in each of the four main domains on a scale of 10
Time Frame: week 16
Population: FAS
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 6 (20.0)

10. Secondary Outcome: Change in Serum Concentration of Secukinumab
Description: The assessment of pre dose concentration of secukinumab in Japanese AS patients
  An enzyme-linked immunosorbent assay (ELISA) method will be used for bioanalytical analysis of secukinumab in serum, with an anticipated lower limit of quantification (LLOQ) of 80 ng/mL.
Time Frame: Baseline, weeks 4, 16, 24, 52, 60
Population: FAS
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
μg/mL
  week 4: number analyzed (Participants) | 28
  week 4 | 51.3 (15.35)
  week 16: number analyzed (Participants) | 29
  week 16 | 25.0 (10.19)
  week 24: number analyzed (Participants) | 27
  week 24 | 22.2 (8.96)
  week 52: number analyzed (Participants) | 24
  week 52 | 21.1 (6.08)
  week 60: number analyzed (Participants) | 23
  week 60 | 6.2 (3.61)

11. Secondary Outcome: Number of Participants With Immunogenicity Against Secukinumab
Description: Concentration of anti-secukinumab antibodies
  Assessment of immunogenicity against secukinumab by concentration of anti-secukinumab antibodies at pre-dose.
  An electrochemiluminescence method was used for the detection of potential anti-secukinumab antibody formation.
Time Frame: week 60
Population: The safety set included all patients who took at least one dose of study treatment during the treatment periods.
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants | 0

12. Secondary Outcome: Number of Participants With Newly Occurring or Worsening Hematology Abnormalities Based on CTCAE Grade, Blood
Description: Common Terminology Criteria for Adverse Events (CTCAE) Grades 1-5 refer to severity of the AE:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL)*.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE.
  *Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
  **Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.
Time Frame: week 60
Population: The safety set included all patients who took at least one dose of study treatment during the treatment periods.
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants
  Hemoglobin (g/L) <LLN - 100 g/L (Grade1): number analyzed (Participants) | 22
  Hemoglobin (g/L) <LLN - 100 g/L (Grade1) | 6
  Hemoglobin (g/L) <100 - 80 g/L (Grade2) | 0
  Hemoglobin (g/L) < 80g/L (Grade3) | 0
  Lymphocytes (10E9/L) <LLN - 0.8 × 10e9/L (Grade1): number analyzed (Participants) | 29
  Lymphocytes (10E9/L) <LLN - 0.8 × 10e9/L (Grade1) | 2
  Lymphocytes (10E9/L) <0.8 - 0.5 × 10e9/L (Grade2) | 1
  Lymphocytes (10E9/L) <0.5 - 0.2 × 10e9/L (Grade3) | 1
  Lymphocytes (10E9/L) <0.2 × 10e9/L (Grade4) | 0
  Neutrophils (10E9/L) < LLN - 1.5 × 10e9/L (Grade1) | 0
  Neutrophils (10E9/L) < 1.5 - 1.0 × 10e9/L (Grade2) | 1
  Neutrophils (10E9/L) < 1.0 - 0.5 × 10e9/L (Grade3) | 0
  Neutrophils (10E9/L) < 0.5 × 10e9/L (Grade4) | 0
  Platelets (10E9/L) <LLN - 75.0 ×10e9/L (Grade1) | 3
  Platelets (10E9/L) <75.0 - 50.0 ×10e9/L (Grade2) | 0
  Platelets (10E9/L) <50.0 - 25.0 ×10e9/L (Grade3) | 0
  Platelets (10E9/L), Blood <25.0 ×10e9/L (Grade4) | 0
  Leukocytes (10E9/L) <LLN - 3.0 × 10e9/L (Grade1) | 0
  Leukocytes (10E9/L) <3.0 - 2.0 × 10e9/L (Grade2) | 1
  Leukocytes (10E9/L) <2.0 - 1.0 × 10e9/L (Grade3) | 0
  Leukocytes (10E9/L) <1.0 × 10e9/L (Grade4) | 0

13. Secondary Outcome: Number of Participants With Newly Occurring or Worsening Chemistry Abnormalities Based on CTCAE Grade
Description: Common Terminology Criteria for Adverse Events (CTCAE) Grades 1-5 refer to severity of the AE:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL)*.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE.
  *Instrumental ADL include preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
  **Self care ADL include bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.
Time Frame: week 60
Population: safety set
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants
  Alkaline Phosphatase (U/L), Serum (Grade1): number analyzed (Participants) | 21
  Alkaline Phosphatase (U/L), Serum (Grade1) | 3
  Alkaline Phosphatase (U/L), Serum (Grade2) | 0
  Alkaline Phosphatase (U/L), Serum (Grade3) | 0
  Alkaline Phosphatase (U/L), Serum (Grade4) | 0
  Alanine Aminotransferase (U/L), Serum (Grade1): number analyzed (Participants) | 28
  Alanine Aminotransferase (U/L), Serum (Grade1) | 3
  Alanine Aminotransferase (U/L), Serum (Grade2) | 0
  Alanine Aminotransferase (U/L), Serum (Grade3) | 0
  Alanine Aminotransferase (U/L), Serum (Grade4) | 0
  Aspartate Aminotransferase (U/L), Serum (Grade1): number analyzed (Participants) | 29
  Aspartate Aminotransferase (U/L), Serum (Grade1) | 4
  Aspartate Aminotransferase (U/L), Serum (Grade2) | 0
  Aspartate Aminotransferase (U/L), Serum (Grade3) | 0
  Aspartate Aminotransferase (U/L), Serum (Grade4) | 0
  Bilirubin (umol/L), Serum (Grade1): number analyzed (Participants) | 29
  Bilirubin (umol/L), Serum (Grade1) | 2
  Bilirubin (umol/L), Serum (Grade2) | 1
  Bilirubin (umol/L), Serum (Grade3) | 0
  Bilirubin (umol/L), Serum (Grade4) | 0
  Cholesterol (mmol/L), Serum (Grade1) Serum: number analyzed (Participants) | 25
  Cholesterol (mmol/L), Serum (Grade1) Serum | 4
  Cholesterol (mmol/L), Serum (Grade2) | 0
  Cholesterol (mmol/L), Serum (Grade3) | 0
  Cholesterol (mmol/L), Serum (Grade4) | 0
  Creatinine (umol/L), Plasma/Serum (Grade1) | 1
  Creatinine (umol/L), Plasma/Serum (Grade2) | 0
  Creatinine (umol/L), Plasma/Serum (Grade3) | 0
  Creatinine (umol/L), Plasma/Serum (Grade4) Serum | 0
  Gamma Glutamyl Transferase (U/L), Serum (Grade1): number analyzed (Participants) | 27
  Gamma Glutamyl Transferase (U/L), Serum (Grade1) | 1
  Gamma Glutamyl Transferase (U/L), Serum (Grade2) | 0
  Gamma Glutamyl Transferase (U/L), Serum (Grade3) | 0
  Gamma Glutamyl Transferase (U/L), Serum (Grade4) | 0
  Glucose Decreased (mmol/L), Plasma (Grade1): number analyzed (Participants) | 29
  Glucose Decreased (mmol/L), Plasma (Grade1) | 0
  Glucose Decreased (mmol/L), Plasma (Grade2) | 0
  Glucose Decreased (mmol/L), Plasma (Grade3) | 0
  Glucose Decreased (mmol/L), Plasma (Grade4) | 0
  Glucose Increased (mmol/L), Plasma (Grade1): number analyzed (Participants) | 26
  Glucose Increased (mmol/L), Plasma (Grade1) | 12
  Glucose Increased (mmol/L), Plasma (Grade2): number analyzed (Participants) | 29
  Glucose Increased (mmol/L), Plasma (Grade2) | 3
  Glucose Increased (mmol/L), Plasma (Grade3) | 1
  Glucose Increased (mmol/L), Plasma (Grade4) | 0
  Triglycerides (mmol/L), Plasma/Serum (Grade1): number analyzed (Participants) | 28
  Triglycerides (mmol/L), Plasma/Serum (Grade1) | 9
  Triglycerides (mmol/L), Plasma/Serum (Grade2): number analyzed (Participants) | 29
  Triglycerides (mmol/L), Plasma/Serum (Grade2) | 1
  Triglycerides (mmol/L), Plasma/Serum (Grade3) | 0
  Triglycerides (mmol/L), Plasma/Serum (Grade4) | 0

14. Secondary Outcome: Participants With Newly Occurring or Worsening Liver Enzyme Abnormalities
Description: During the entire safety reporting period, mean values of each liver enzyme parameter stayed within the normal range and were comparable to the baseline values
  ALP=Alkaline phosphatase ALT=Alanine aminotransferase AST=Aspartate aminotransferase TBL=Total bilirubin ULN=Upper Limit Normal
Time Frame: week 60
Population: safety set
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants
  ALT > 3 × ULN | 0
  ALT > 5 × ULN | 0
  ALT > 8 × ULN | 0
  ALT > 10 × ULN | 0
  ALT > 20 × ULN | 0
  AST > 3 × ULN | 0
  AST > 5 × ULN | 0
  AST > 8 × ULN | 0
  AST > 10 × ULN | 0
  AST > 20 × ULN | 0
  ALT or AST > 3 × ULN | 0
  ALT or AST > 5 × ULN | 0
  ALT or AST > 8 × ULN | 0
  ALT or AST > 10 × ULN | 0
  ALT or AST > 20 × ULN | 0
  TBL > 1.5 × ULN | 1
  TBL > 2 × ULN | 0
  TBL > 3 × ULN | 0
  ALP > 2 × ULN | 0
  ALP > 3 × ULN | 0
  ALP > 5 × ULN | 0
  ALT or AST > 3 × ULN & TBL > 2 × ULN | 0
  ALT or AST > 5 × ULN & TBL > 2 × ULN | 0
  ALT or AST > 8 × ULN & TBL > 2 × ULN | 0
  ALT or AST > 10 × ULN & TBL > 2 × ULN | 0
  ALP > 3 × ULN & TBL > 2 × ULN | 0
  ALP > 5 × ULN & TBL > 2 × ULN | 0
  ALT or AST> 3 × ULN & TBL> 2 × ULN & ALP <2 × ULN | 0

15. Secondary Outcome: Number of Participants With Newly Occurring or Worsening Lipid Parameters Abnormalities
Description: During the entire safety reporting period, mean values of each lipid parameter stayed within the normal range and were comparable to the baseline values
Time Frame: week 60
Population: safety set
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants
  HDL: ≤ LLN: number analyzed (Participants) | 26
  HDL: ≤ LLN | 5
  HDL: < 0.8 × LLN: number analyzed (Participants) | 29
  HDL: < 0.8 × LLN | 1
  LDL: ≥ ULN: number analyzed (Participants) | 23
  LDL: ≥ ULN | 1
  LDL: > 1.5 × ULN | 0
  LDL: > 2.5 × ULN | 0
  Cholesterol: ≥ ULN: number analyzed (Participants) | 25
  Cholesterol: ≥ ULN | 4
  Cholesterol: > 1.5 × ULN | 0
  Cholesterol: > 2.5 × ULN | 0
  Triglycerides: ≥ ULN: number analyzed (Participants) | 27
  Triglycerides: ≥ ULN | 8
  Triglycerides: > 1.5 × ULN: number analyzed (Participants) | 29
  Triglycerides: > 1.5 × ULN | 4
  Triglycerides: > 2.5 × ULN | 0

16. Secondary Outcome: Participants With Newly Occurring Notable Abnormalities in Vital Signs
Description: Sitting Pulse (bpm) High only (> 100 bpm) Low only (< 60 bpm) Low and High (< 60 bpm and > 100 bpm)
  Sitting Diastolic Blood Pressure (BP) (mmHg) High only (≥ 90 mmHg) Low only (< 60 mmHg) Low and High (< 60 mmHg and ≥ 90 mmHg)
  Sitting Systolic Blood Pressure (mmHg) High only (≥ 140 mmHg) Low only (< 90 mmHg) Low and High (< 90 mmHg and ≥ 140 mmHg)
Time Frame: week 60
Population: safety set
Measure: Number; unit: participants
Arm/Group | Secukinumab 150mg
Number analyzed (Participants) | 30
participants
  Sitting Pulse (bpm) High only | 2
  Sitting Pulse (bpm) Low only: number analyzed (Participants) | 28
  Sitting Pulse (bpm) Low only | 5
  Sitting Pulse (bpm) Low and High: number analyzed (Participants) | 28
  Sitting Pulse (bpm) Low and High | 0
  Sitting Diastolic BP (mmHg), High only: number analyzed (Participants) | 26
  Sitting Diastolic BP (mmHg), High only | 8
  Sitting Diastolic BP (mmHg), Low only | 5
  Sitting Diastolic BP (mmHg), Low and high: number analyzed (Participants) | 26
  Sitting Diastolic BP (mmHg), Low and high | 0
  Sitting Systolic BP (mmHg) High only: number analyzed (Participants) | 27
  Sitting Systolic BP (mmHg) High only | 12
  Sitting Systolic BP (mmHg) Low only | 0
  Sitting Systolic BP (mmHg) Low and High: number analyzed (Participants) | 27
  Sitting Systolic BP (mmHg) Low and High | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 60 weeks. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 60 weeks
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 60 weeks
Groups:
- AIN457 150mg: A screening (SCR) epoch ran 4-10 weeks before baseline (BSL) and was used to assess eligibility followed by 52 weeks of treatment. The treatment periods consisted of Treatment period 1 (BSL to Week 24) and Treatment period 2 (Week 24 to Week 52). After Week 52 there was a post-treatment follow-up until Week 60. A follow-up visit was done at 12 weeks after last study treatment administration for all patients, regardless of whether they completed the entire study as planned (Week 60) or discontinued prematurely.
Arm/Group | AIN457 150mg
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150mg (N=30)
Coronary artery occlusion (Cardiac disorders) | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150mg (N=30)
Leukopenia (Blood and lymphatic system disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 3
Infected dermal cyst (Infections and infestations) | 2
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 15
Pharyngitis (Infections and infestations) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
This single arm study has no comparator and therefore no statistical test for comparison was planned for the outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-11-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT02750592/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT02750592/SAP_001.pdf